CLINICAL TRIAL: NCT02525523
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of the Safety and Efficacy of Topical Alicaforsen Enema in Subjects With Active, Chronic, Antibiotic Refractory Primary Idiopathic Pouchitis
Brief Title: Efficacy of Alicaforsen in Pouchitis Patients Who Have Failed to Respond to at Least One Course of Antibiotics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Atlantic Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACH UCP-301
Record Dates: First submitted 2015-08-14; First posted 2015-08-17 (Estimated); Results first posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Pouchitis
MeSH Terms: conditions — Pouchitis | interventions — alicaforsen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Alicaforsen (Experimental): Alicaforsen enema, 240mg once daily for 6 weeks
  Interventions: Drug: Alicaforsen
- Placebo (Placebo Comparator): Placebo enema, once daily for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alicaforsen
  Arms: Alicaforsen
Drug: Placebo
  Arms: Placebo

SUMMARY:
A Phase III, multi-centre, double-blind randomised controlled trial in subjects with chronic antibiotic refractory pouchitis.

Subjects will undertake a <2 week screening period to provide baseline data and be assessed for eligibility. At the Baseline visit (Day 1) eligible subjects will be randomised on a 1:1 basis to either a) 240 mg alicaforsen enema or b) matching placebo.

Study drug will be administered once nightly (on going to bed) up to and including week 6. Following the Day 1 Visit, subjects will return to the clinic for safety and efficacy assessments at Week 3, 6, 10, 18 and 26.

Subjects may receive certain permitted medications as per Entry Criteria, which must remain at stable doses throughout the trial. Introduction of any new medication for pouchitis, or a dose change to an existing concomitant medication for pouchitis, other than those detailed in the protocol, will not be permitted.

Clinical symptoms associated with pouchitis will be recorded daily by the patient in a diary card.

Subjects will undergo endoscopic examination of their pouch (during Screening, and at Weeks 6 and 10). Where technically feasible, each endoscopy will provide at least one biopsy sample for histopathology.

In addition to endoscopic, histopathologic and symptomatic assessments, Quality of Life will be assessed.

Bloods for routine assessment, including haematology and biochemistry will be taken. Bloods and stool samples will be collected to evaluate relevant biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent;
2. Male or female subjects, 18 years of age who have undergone an IPAA for UC
3. History of pouchitis
4. Overall PDAI score > 7
5. Must have Chronic Antibiotic Refractory Pouchitis

Exclusion Criteria:

1. Lack of effective contraception
2. Women who are pregnant or breastfeeding;
3. Strong analgesia NSAID use
4. Change in dose of the following permitted meds during screening and study: oral 5-aminosalicylate (5 ASA), Oral steroids,, Immunosuppressant therapy.
5. Rectal products
6. Biological agents: Anti-tumour necrosis factor (anti - TNF) therapy and / or vedolizumab; are not permitted within 8 weeks of the Screening Visit.
7. All other agents targeted to pouchitis, including experimental agents, must have been discontinued at least 8 weeks prior to the Screening Visit, or for a period equivalent to 5 half-lives (t½) of the agent (whichever is longer)
8. Anal sphincter dysfunction
9. Infections to cytomegalovirus or Clostridium Difficile
10. Other GI pathology (inc. intestinal malabsorption, pancreatic maldigestion etc) and differential diagnoses
11. Clinically significant and/or persistent illness; which in the investigators opinion, would exclude entry into the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2015-12-03 (Actual); Primary Completion 2018-07-09 (Actual); Study Completion 2018-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Dunk, Study Director — Atlantic Pharmaceuticals
Locations (41):
- United States (12):
  - Site Reference ID/Investigator# 1008, La Jolla, California
  - Site Reference ID/Investigator # 1005, Los Angeles, California
  - Site Reference ID/Investigator#1011, Stanford, California
  - Site Reference ID/Investigator#1012, Atlanta, Georgia
  - Site Reference ID/Investigator# 1010, Chicago, Illinois
  - Site Reference ID/Investigator# 1001, Rochester, Minnesota
  - Site Reference ID/Investigator# 1003, Great Neck, New York
  - Site Reference ID/Investigator# 1006, New York, New York
  - Site Reference ID/Investigator# 1009, New York, New York
  - Site Reference ID/Investigator# 1004, Cleveland, Ohio
  - Site Reference ID/Investigator# 1002, Oklahoma City, Oklahoma
  - Site Reference ID/Investigator# 1007, Seattle, Washington
- Belgium (3):
  - Site Reference ID/Investigator# 0103, Brussels
  - Site Reference ID/Investigator# 0102, Ghent
  - Site Reference ID/Investigator# 0101, Leuven
- Canada (5):
  - Site Reference ID/Investigator# 0205, Calgary, Alberta
  - Site Reference ID/Investigator# 0201, Edmonton, Alberta
  - Site Reference ID/Investigator# 0204, Vancouver, British Columbia
  - Site Reference ID/Investigator# 0202, London, Ontario
  - Site Reference ID/Investigator# 0203, Toronto, Ontario
- France (4):
  - Site Reference ID/Investigator# 0403, Lille
  - Site Reference ID/Investigator# 0402, Nice
  - Site Reference ID/Investigator# 0401, Saint-Etienne
  - Site Reference ID/Investigator# 0404, Toulouse
- Ireland (2):
  - Site Reference ID/Investigator# 0601, Dublin
  - Site Reference ID/Investigator# 0602, Dublin
- Site Reference ID/Investigator# 0701, Tel Aviv, Israel
- Italy (4):
  - Site Reference ID/Investigator# 0801, Bologna
  - Site Reference ID/Investigator# 0804, Rome
  - Site Reference ID/Investigator# 0803, Rome
  - Site Reference ID/Investigator# 0802, Rozzano
- Netherlands (2):
  - Site Reference ID/Investigator# 0901, Amsterdam
  - Site Reference ID/Investigator# 0902, Nijmegen
- Switzerland (2):
  - Site Reference ID/Investigator# 0302, Bern
  - Site Reference ID/Investigator# 0301, Zurich
- United Kingdom (6):
  - Site Reference ID/Investigator# 0504, Harrow, Middlesex
  - Site Reference ID/Investigator# 0501, Nottingham, Nottinghamshire
  - Site Reference ID/Investigator# 0503, Coventry, Warwickshire
  - Site Reference ID/Investigator# 0506, Birmingham
  - Site Reference ID/Investigator# 0502, London
  - Site Reference ID/Investigator# 0505, London

RESULTS

PARTICIPANT FLOW:
Groups:
- Alicaforsen: Alicaforsen enema, 240mg once daily for 6 weeks
  Alicaforsen
- Placebo: Placebo enema, once daily for 6 weeks
  Placebo
Period: Overall Study
Arm/Group | Alicaforsen | Placebo
Started | 69 | 69
Completed | 46 | 44
Not Completed | 23 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alicaforsen | Placebo | Total
Number analyzed (Participants) | 69 | 69 | 138
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 65 | 66 | 131
  >=65 years | 4 | 3 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 28 | 58
  Male | 39 | 41 | 80
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 5 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 62 | 54 | 116
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 10 | 15

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Endoscopic Remission
Description: The group of patients with an improvement in their endoscopic score between screening and week 10 as shown by an reduced modified MAYO score. Remission is defined as absence of friability and ulceration, represented by a score of ≤1.
Time Frame: Week 10
Measure: Count of Participants; unit: Participants
Arm/Group | Alicaforsen | Placebo
Number analyzed (Participants) | 65 | 61
Participants | 3 | 3

2. Primary Outcome: Proportion of Patients With a Reduction in Relative Stool Frequency
Description: Group of patients with a lowering of stool frequency from baseline to week 10, where the subject's stool frequency is represented by a MAYO subscore of ≤1 at week 10.
Time Frame: Week 10
Measure: Count of Participants; unit: Participants
Arm/Group | Alicaforsen | Placebo
Number analyzed (Participants) | 65 | 61
Participants | 22 | 16

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Alicaforsen | Placebo
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/69
Serious Adverse Events (participants affected / at risk) | 4/69 | 2/69
Other Adverse Events (participants affected / at risk) | 19/69 | 20/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alicaforsen (N=69) | Placebo (N=69)
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Anal Absess (Infections and infestations) | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Facial Paralysis (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alicaforsen (N=69) | Placebo (N=69)
Abdominal pain (Gastrointestinal disorders) | 2 | 7
Pouchitis (Gastrointestinal disorders) | 4 | 5
Anorectal discomfort (Gastrointestinal disorders) | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 4 | 1
Nasopharyngitis (Infections and infestations) | 6 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-08-19): https://cdn.clinicaltrials.gov/large-docs/23/NCT02525523/Prot_000.pdf
  • Statistical Analysis Plan (2016-08-19): https://cdn.clinicaltrials.gov/large-docs/23/NCT02525523/SAP_001.pdf